CLINICAL TRIAL: NCT02457819
Title: An Open-label, Flexibly-dosed, 26-Week Extension Safety Study of Dasotraline in Children and Adolescents With Attention Deficit Hyperactivity Disorder (ADHD)
Brief Title: Dasotraline Pediatric Extension Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SEP360-310
Record Dates: First submitted 2015-05-20; First posted 2015-05-29 (Estimated); Results first posted 2020-01-18 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — 4-(3,4-dichlorophenyl)-1,2,3,4-tetrahydronaphthalen-1-amine

STUDY DESIGN:
Masking Description: Open label
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dasotraline (Experimental): Dasotraline 2, 4, 6 mg
  Interventions: Drug: Dasotraline

INTERVENTIONS:
Drug: Dasotraline — Dasotraline 2 mg, 4 mg, 6 mg, once daily, flexibly dosed

SUMMARY:
This is an open label 26 week extension study for subjects who completed SEP360-202.

DETAILED DESCRIPTION:
This is an open-label, flexibly-dosed, 26 week extension study in children and adolescents with ADHD who have completed 6 weeks of double-blind treatment in the core study (SEP360 202). This study will evaluate the long-term safety and tolerability of dasotraline in this population.

ELIGIBILITY:
Inclusion Criteria:

* At least one of the subject's parent/legal guardian must give written informed consent, including privacy authorization, prior to study participation. The subject will complete an informed assent prior to study participation.
* Subject and subject's parent/legal guardian are judged by the investigator to be willing and able to comply with the study procedures and visit schedules.
* Subject has completed all required assessments for Week 6 of the core study.
* Subject has not taken any medication other than the study drug for the purpose of controlling ADHD symptoms during the core study.
* Subject, if female, must not be pregnant or breastfeeding.
* Female subject: must be unable to become pregnant (eg, premenarchal, surgically sterile, etc);

-OR-

* practice true abstinence (consistent with lifestyle) and must agree to remain abstinent from signing informed consent/assent to at least 14 days after the last dose of study drug has been taken; -OR-
* is sexually active and willing to use a medically effective method of birth control from signing informed consent/assent to at least 14 days after the last dose of study drug has been taken.
* Male subject must be willing to remain sexually abstinent (consistent with lifestyle) or use an effective method of birth control, from signing informed consent/assent to at least 14 days after the last dose of study drug has been taken.
* Any subject whose weight is less than or equal to 21 kg at the OL Baseline visit should be discussed with the medical monitor prior to enrollment.
* Subject and subject's parent/legal guardian must be able to fully comprehend the informed consent/assent form (as applicable), understand all study procedures, and be able to communicate satisfactorily with the Investigator and study coordinator.

Exclusion Criteria:

* -Subject is considered by the investigator to be at imminent risk of suicide, injury to self or to others, or damage to property.
* Subject answers "yes" to "Suicidal Ideation" item 4 (active suicidal ideation with some intent to act, without specific plan) or item 5 (active suicidal ideation with specific plan and intent) for any lifetime history on the C SSRS Children's "Since Last Visit" assessment at OL Baseline.
* Subject has a clinically significant abnormality including physical examination, vital signs, ECG, or laboratory tests that the investigator in consultation with the medical monitor considers to be inappropriate to allow participation in the study.
* Subject has a positive urine drug screen (UDS) or breath alcohol test at OL Baseline.
* Subject or parents/legal guardian has commitments during the study that would interfere with attending study visits.
* Subject is at high risk of non-compliance in the investigator's opinion.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 237 (Actual)
Dates: Start 2015-06-30 (Actual); Primary Completion 2017-02-02 (Actual); Study Completion 2017-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dasotraline Medical Director, Study Director — Sumitomo Pharma America, Inc.
Locations (36):
- United States (36):
  - Harmonex Neuroscience Research, Inc, Dothan, Alabama
  - ProScience Research Group, Culver City, California
  - Elite Clinical Trials, Inc., Wildomar, California
  - MCB Clinical Research Centers, LLC, Colorado Springs, Colorado
  - Sarkis Clinical Trials, Gainesville, Florida
  - Indago Research Health Center, Inc., Hialeah, Florida
  - Clinical Neuroscience Solutions, Inc, Jacksonville, Florida
  - Florida Clinical Research Center, LLC, Maitland, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Miami Research Associates, LLC, South Miami, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - iResearch Atlanta, LLC, Decatur, Georgia
  - Capstone Clinical Research, Libertyville, Illinois
  - Baber Research Group, Inc., Naperville, Illinois
  - Goldpoint Clinical Research, LLC., Indianapolis, Indiana
  - Pedia Research,LLC, Newburgh, Indiana
  - Psychiatric Associates, Overland Park, Kansas
  - Pedia Research,LLC, Owensboro, Kentucky
  - Neurobehavioral Medicine Group, Clinical Trials Division, Bloomfield Hills, Michigan
  - Clinical Trials group at the Rochester Center for Behavioral Medicine, Rochester Hills, Michigan
  - St. Charles Psychiatric Associates - Midwest Research Group, Saint Charles, Missouri
  - Center for Psychiatry and Behavioral Medicine, Inc., Las Vegas, Nevada
  - Pharmaceutical Research Associates, Inc., Marlton, New Jersey
  - Richarmond Behavioral Associates, Staten Island, New York
  - University of Cincinnati/Department of Psychiatry and Behavioral Neuroscience, Cincinnati, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Cutting Edge Research Group, Oklahoma City, Oklahoma
  - Cyn3rgy Research, Gresham, Oregon
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - BioBehavioral Research of Austin P.C., Austin, Texas
  - Bayou City Research, Ltd., Houston, Texas
  - Houston Clinical Trials, LLC, Houston, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Road Runner Research, Ltd., San Antonio, Texas
  - Family Psychiatry of the Woodlands, The Woodlands, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Dasotraline: Dasotraline 2, 4, 6 mg, flexibly dosed
Period: Overall Study
Arm/Group | Dasotraline
Started | 237
Safety Population | 236
Completed | 138
Not Completed | 99
Not completed — reason not given | 8
Not completed — Withdrawal by Subject | 24
Not completed — Protocol Violation | 1
Not completed — non compliance with study drug | 4
Not completed — Lost to Follow-up | 10
Not completed — Lack of Efficacy | 19
Not completed — Adverse Event | 33

BASELINE CHARACTERISTICS:
Arm/Group | Dasotraline
Number analyzed (Participants) | 236
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 236
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76
  Male | 160
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 37
  Not Hispanic or Latino | 199
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 71
  White | 146
  More than one race | 7
  Unknown or Not Reported | 9
Region of Enrollment [Number; unit: participants] — United States
  participants
    United States | 236

OUTCOME MEASURES:

1. Primary Outcome: The Incidence of Overall Adverse Events, AEs , Serious Adverse Envents,(or SAEs), and AEs (or SAEs) Leading to Discontinuation
Description: Overall adverse events, AEs , serious adverse envents,(or SAEs), and AEs (or SAEs) leading to discontinuation.
Time Frame: 26 Weeks
Population: safety population
Measure: Number; unit: adverse events
Arm/Group | Dasotraline
Number analyzed (Participants) | 236
adverse events
  Subjects with any TEAE | 144
  Subjects with any TEAE leading to discontinuation | 30
  Subjects with any serious TEAE | 3
  Subjects with any serious treatment-related TEAE | 1
  treatment-related TEAE leading to discontinuation | 1

2. Secondary Outcome: Change From Baseline, in Attention Deficit Hyperactivity Disorder Rating Scale, Version IV, Home Version, (ADHD RS IV HV) Total Score.
Description: The ADHD RS-IV HV is a validated scale that consists of 18 items designed to reflect current symptomatology of ADHD based on Diagnostic and Statistical Manual for Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) criteria and is also consistent with DSM-5 criteria.
  Each item is scored from a range of zero (reflecting no symptoms) to 3 (reflecting severe symptoms) with total scores ranging from zero to 54. The 18 items may be grouped into 2 subscales: hyperactivity/impulsivity (even number items 2 through 18) and inattentiveness (odd number items 1 through 17).
Time Frame: 26 Weeks
Population: safety population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dasotraline
Number analyzed (Participants) | 138
units on a scale | -7.1 (10.19)

3. Secondary Outcome: Change From Baseline, in Clinical Global Impression-Severity of Illness (CGI S) Score.
Description: The CGI-S scale, modified captures the clinician's rating of observed and reported ADHD symptoms, behavior, and function over the past 7 days. The CGI-S is rated on the following 7-point scale: 1 = normal, not at all ill; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; and 7 = among the most extremely ill subjects.
Time Frame: 26 weeks
Population: safety population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dasotraline
Number analyzed (Participants) | 139
units on a scale | -0.6 (1.11)

ADVERSE EVENTS:
Time Frame: 26 weeks
Arm/Group | Dasotraline
All-Cause Mortality (participants affected / at risk) | 0/236
Serious Adverse Events (participants affected / at risk) | 3/236
Other Adverse Events (participants affected / at risk) | 94/236
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dasotraline (N=236)
Pyelonephritis (Infections and infestations) | 1 (1)
Psychomotor hyperactivity (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Panic attack (Product Issues) | 1 (1)
Substance-induced psychotic disorder (Psychiatric disorders) | 1 (1)
Suicidal ideatin (Psychiatric disorders) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dasotraline (N=236)
Weight decreased (Investigations) | 29 (30)
Decreased apppetite (Metabolism and nutrition disorders) | 49 (56)
Headache (Nervous system disorders) | 26 (31)
Anxiety (Nervous system disorders) | 13 (15)
Initial insomnia (Nervous system disorders) | 26 (30)
Irritability (Nervous system disorders) | 20 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In the event the Study is part of a multi-center study, the first publication of the results of the Study shall be made in conjunction with the results of other participating study sites as a multi-center publication; provided however, if a multi-center publication is not forthcoming within twenty-four (24) months following completion of the Study at all sites, Institution and Investigator shall be free to publish.

DOCUMENTS (2):
  • Study Protocol (2016-01-20): https://cdn.clinicaltrials.gov/large-docs/19/NCT02457819/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-09): https://cdn.clinicaltrials.gov/large-docs/19/NCT02457819/SAP_001.pdf